CLINICAL TRIAL: NCT06233864
Title: A Phase II Clinical Study of the Treatment of Disitamab Vedotin（RC48) in Patients With Locally Advanced or Metastatic Pancreatic Cancer Expressing HER2
Brief Title: A Study of the Treatment of Disitamab Vedotin in Patients With Locally Advanced or Metastatic Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dong sheng Zhang, PHD, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M01-RC48
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — disitamab vedotin; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disitamab Vedotin combined with Gemcitabine，2L (Experimental): Disitamab Vedotin 2.5 mg/kg，iv，Q3W; Gemcitabine 1g/m2，iv，d1, d8 Q3W; Disitamab Vedotin+Gemcitabine is used as second-line treatment for HER2-expressive patients who have failed first-line gemcitabine-free regimen or are intolerant to gemcitabine-containing regimen.
  Interventions: Drug: Disitamab Vedotin; Drug: Gemcitabine
- Disitamab Vedotin，3L (Experimental): Disitamab Vedotin 2.5 mg/kg，iv，Q3W; Disitamab Vedotin in HER2-expressive patients who have failed at second-line standard treatment or are intolerant
  Interventions: Drug: Disitamab Vedotin

INTERVENTIONS:
Drug: Disitamab Vedotin — Disitamab Vedotin
  Other Names: RC48
Drug: Gemcitabine — Gemcitabine
  Arms: Disitamab Vedotin combined with Gemcitabine，2L

SUMMARY:
This is a phase 2 clinical study,to explore the efficacy and safety of Disitamab Vedotin in patients with locally advanced or metastatic pancreatic cancer expressing HER2.

DETAILED DESCRIPTION:
63 patients with locally advanced or metastatic pancreatic cancer will participate in this study. HER2 expression in locally advanced or metastatic pancreatic cancer patients is defined as the expression of HER2 in tumor tissues detected by immunohistochemistry (IHC) as IHC 1+, 2+, or 3+. The arm 1 recruits 43 patients and the arm 2 recruits 20 patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18 (inclusive) or above, regardless of gender.
* 2. histologically or cytologically confirmed patients with locally advanced or metastatic pancreatic cancer who cannot undergo radical surgery
* 3. HER2 expressing(Immunohistochemical IHC 1+,2+ or 3+)
* 4. Number of treatment lines: Cohort 1: Prior first-line gemcitabine-free regimen or intolerant to gemcitabine-containing regimen; Cohort 2: Previous treatment with second-line standard or intolerance
* 5. Patients who have previously received neoadjuvant chemotherapy, adjuvant chemotherapy, radiotherapy or chemoradiotherapy for the purpose of curing non-metastatic disease must have a disease-free interval of 6 months from the last chemotherapy and/or radiotherapy to the random date
* 6. There is at least one measurable lesion that meets the definition of the RECIST 1.1 standard at baseline.
* 7. ECOG fitness status score: 0 or 1 point.
* 8. Estimated survival time ≥ 3 months.
* 9. Adequate organ function.
* 10. Male and female participants are eligible to participate if they agree to the contraception use as per study protocol.
* 11. Voluntary agreement to provide written informed consent.

Exclusion Criteria:

* 1. Central nervous system metastasis or meningeal metastasis with clinical symptoms.
* 2. Have a history of autoimmune diseases, immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation.
* 3. Active hepatitis B (hepatitis B virus titer>1000 copies/ml or 200 IU/ml); Hepatitis C virus and syphilis infection.
* 4. Have undergone major organ surgery (excluding puncture biopsy) or have experienced significant trauma within 3 weeks before the first use of the study drug.
* 5. Known hypersensitivity or intolerance to any component of the study protocol drug or its excipients.
* 6. Strong inducers and inhibitors of P-gp, a strong or moderate inducer of CYP3A4, used within 14 days prior to the first use of the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-04-17 (Estimated); Primary Completion 2025-04-17 (Estimated); Study Completion 2026-04-17 (Estimated)

PRIMARY OUTCOMES:
Object Response Rate, ORR | up to 12 months
  Defined as the percentage of participants with a complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Disease Control Rate, DCR | up to 12 months
  Defined as the proportion of participants who have a complete response (CR), partial response (PR) or standard disease (SD) as assessed by investigator according to RECIST 1.1
Progress Free Survival, PFS | up to 12 months
  Defined as time from randomization until progression per RECIST 1.1 as assessed by investigator, or death due to any cause.
Over Survival, OS | up to 12 months
  Defined as time from randomization until the date of death due to any cause.
Adverse Events (AE) | up to 12 months
  NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Dong sheng Zhang, PhD, Principal Investigator — Sun Yat-sen University Cancer Center, State Key Laboratory of Oncology in South China